CLINICAL TRIAL: NCT07297238
Title: Therapeutic Efficacy of GLP-1 on Intestinal Barrier Function in Patients With Short Bowel Syndrome and Intestinal Failure: A Preliminary Randomized Controlled Trial
Brief Title: Effect of GLP-1 on Intestinal Barrier Function in SBS-IF Patients: A Preliminary Exploration.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Wang Xinying, Prof, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-09-17
Record Dates: First submitted 2025-09-19; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Short Bowel Syndrome (SBS); Intestinal Failure
Keywords: GLP-1; short bowel syndrome; intestinal failure; Intestinal Barrier Function
MeSH Terms: conditions — Short Bowel Syndrome; Intestinal Failure | interventions — Glucagon-Like Peptide-1 Receptor Agonists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Participants received semaglutide as a subcutaneous injection (dosage form) at a dose of 0.25 mg (dosage) once weekly (frequency) for 28 days (duration).
  Interventions: Drug: GLP-1 Receptor Agonists
- Control arm (No Intervention): received appearance-matched placebo plus standard care, no additional semaglutide intervention therapy

INTERVENTIONS:
Drug: GLP-1 Receptor Agonists — GLP-1 receptor agonists (semaglutide) are medications that mimic the action of the native human hormone glucagon-like peptide-1 (GLP-1). The recommended dosage is 0.25 mg administered subcutaneously once weekly.
  Other Names: GLP-1RAs
  Arms: Experimental arm

SUMMARY:
Eligible patients were randomized into two groups: the GLP-1 group and the control group. The control group received a placebo along with standard care, without any additional GLP-1-based intervention. The GLP-1 group, in addition to standard care, received a subcutaneous injection of a GLP-1 analog (semaglutide injection) strictly according to the drug manufacturer's instructions. The initial dose of semaglutide was 0.25 mg once weekly. Treatment was continued over a 28-days period. Primary and secondary outcomes will be collected.

DETAILED DESCRIPTION:
Eligible patients with short bowel syndrome and intestinal failure were randomly assigned to one of two groups: the GLP-1 group or the control group. The control group received a placebo along with standard care. The GLP-1 group, in addition to standard care, was administered a GLP-1 analog (semaglutide injection) via subcutaneous injection strictly according to the manufacturer's instructions, with an initial dose of semaglutide of 0.25 mg once weekly. Primary and secondary outcomes will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Participants voluntarily provided written informed consent for this trial;
* Aged 18 to 80 years, inclusive, regardless of gender;
* With stable vital signs;
* Diagnosis of SBS-IF, confirmed by existing medical/surgical records, receiving parenteral nutrition (PN) due to surgical resection of the small intestine (<200 cm from the duodenojejunal flexure), and meeting one of the following criteria:

  * Colon continuity maintained without jejunal/ileal stoma (Type II or III);

    * Presence of a jejunostomy or ileostomy (Type I);
* Expected requirement of PN for more than 4 weeks, with an average PN caloric intake ≥80%;
* Ability to comply with the medication dosing and visit schedule;
* Capacity to accurately describe symptoms, absence of severe infections or respiratory insufficiency, and willingness to cooperate proactively;
* No history of allergic diseases, non-allergic constitution, and no hypersensitivity to any component of semaglutide injection;
* No history of drug abuse;
* Not pregnant or lactating; no pregnancy plans within one month after the trial (applies to both female and male participants);
* No participation in any other drug trials (including the investigational product in this study) within three months prior to enrollment.

Exclusion Criteria:

* Individuals who do not meet the inclusion criteria or are deemed ineligible by the investigator;
* Poor general condition, inability to accurately describe symptoms, presence of severe infection, respiratory insufficiency, or other conditions that may hinder active cooperation;
* History of allergic diseases, allergic constitution, or hypersensitivity to drugs structurally related to the investigational product;
* Patients with malignancy at any site;
* Those with psychiatric disorders, inability to cooperate, or impaired consciousness;
* Patients with contraindications to the investigational drug (including personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2);
* Immunodeficiency, or current use of immunosuppressants or corticosteroids;
* Immediate family members of the sponsor, investigator, or study staff directly involved in the trial;
* Any other condition considered by the investigator as grounds for exclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Serum Biomarkers of Intestinal Barrier Function | the initiation of enrollment and upon completion of the 28-days treatment period
  Serum Citrulline（µmol/L）

SECONDARY OUTCOMES:
Intestinal absorption of nutrients (protein) | the initiation of enrollment and upon completion of the 28-days treatment period
  Intestinal nitrogen balance（Kjeldahl method for total nitrogen intake and excretion）
Intestinal absorption of nutrients (carbohydrate) | the initiation of enrollment and upon completion of the 28-days treatment period
  Fecal carbohydrate（Fecal pH measurement and analysis of fermentable substrates for indirect assessment）
Intestinal absorption of nutrients (fat) | the initiation of enrollment and upon completion of the 28-days treatment period
  Fat excretion rates（van de Kamer method for direct measurement of total fecal fat excretion）
Nutritional status indicator | the initiation of enrollment and upon completion of the 28-days treatment period
  Serum albumin (g/L) level
PN Liberation Rate | the initiation of enrollment and upon completion of the 28-days treatment period
  A 20% reduction in the weekly parenteral nutrition volume from baseline
Quality of life score | the initiation of enrollment and upon completion of the 28-days treatment period
  Quality of life was assessed using the SF-36 score from the date of randomization until the end of the 4-week intervention weeks. SF-36 consists of eight dimensions, each of which is measured on a scale of 0-100, with higher scores indicating a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Xinying Wang, MD, Principal Investigator — Jinling Hospital, China
Locations (1):
- Jinling Hospital, Nanning, China, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kissow H, Hartmann B, Holst JJ, Poulsen SS. Glucagon-like peptide-1 as a treatment for chemotherapy-induced mucositis. Gut. 2013 Dec;62(12):1724-33. doi: 10.1136/gutjnl-2012-303280. Epub 2012 Oct 20. PMID 23086829
- [Background] Bang-Berthelsen CH, Holm TL, Pyke C, Simonsen L, Sokilde R, Pociot F, Heller RS, Folkersen L, Kvist PH, Jackerott M, Fleckner J, Vilien M, Knudsen LB, Heding A, Frederiksen KS. GLP-1 Induces Barrier Protective Expression in Brunner's Glands and Regulates Colonic Inflammation. Inflamm Bowel Dis. 2016 Sep;22(9):2078-97. doi: 10.1097/MIB.0000000000000847. PMID 27542128
- [Background] Zou Z, Wang Z. Liraglutide attenuates intestinal ischemia/reperfusion injury via NF-kappaB and PI3K/Akt pathways in mice. Life Sci. 2022 Nov 15;309:121045. doi: 10.1016/j.lfs.2022.121045. Epub 2022 Oct 4. PMID 36206837
- [Background] Thazhath SS, Marathe CS, Wu T, Chang J, Khoo J, Kuo P, Checklin HL, Bound MJ, Rigda RS, Crouch B, Jones KL, Horowitz M, Rayner CK. The Glucagon-Like Peptide 1 Receptor Agonist Exenatide Inhibits Small Intestinal Motility, Flow, Transit, and Absorption of Glucose in Healthy Subjects and Patients With Type 2 Diabetes: A Randomized Controlled Trial. Diabetes. 2016 Jan;65(1):269-75. doi: 10.2337/db15-0893. Epub 2015 Oct 15. PMID 26470783
- [Background] Madsen KB, Askov-Hansen C, Naimi RM, Brandt CF, Hartmann B, Holst JJ, Mortensen PB, Jeppesen PB. Acute effects of continuous infusions of glucagon-like peptide (GLP)-1, GLP-2 and the combination (GLP-1+GLP-2) on intestinal absorption in short bowel syndrome (SBS) patients. A placebo-controlled study. Regul Pept. 2013 Jun 10;184:30-9. doi: 10.1016/j.regpep.2013.03.025. Epub 2013 Mar 16. PMID 23511332
- [Background] Hvistendahl M, Brandt CF, Tribler S, Naimi RM, Hartmann B, Holst JJ, Rehfeld JF, Hornum M, Andersen JR, Henriksen BM, Brobech Mortensen P, Jeppesen PB. Effect of Liraglutide Treatment on Jejunostomy Output in Patients With Short Bowel Syndrome: An Open-Label Pilot Study. JPEN J Parenter Enteral Nutr. 2018 Jan;42(1):112-121. doi: 10.1177/0148607116672265. Epub 2017 Dec 11. PMID 27875281
- [Background] Pironi L, Arends J, Baxter J, Bozzetti F, Pelaez RB, Cuerda C, Forbes A, Gabe S, Gillanders L, Holst M, Jeppesen PB, Joly F, Kelly D, Klek S, Irtun O, Olde Damink SW, Panisic M, Rasmussen HH, Staun M, Szczepanek K, Van Gossum A, Wanten G, Schneider SM, Shaffer J; Home Artificial Nutrition & Chronic Intestinal Failure; Acute Intestinal Failure Special Interest Groups of ESPEN. ESPEN endorsed recommendations. Definition and classification of intestinal failure in adults. Clin Nutr. 2015 Apr;34(2):171-80. doi: 10.1016/j.clnu.2014.08.017. Epub 2014 Sep 21. PMID 25311444
- [Background] Doola R, Greer RM, Hurford R, Flatley C, Forbes JM, Todd AS, Joyce CJ, Sturgess DJ. Glycaemic variability and its association with enteral and parenteral nutrition in critically ill ventilated patients. Clin Nutr. 2019 Aug;38(4):1707-1712. doi: 10.1016/j.clnu.2018.08.001. Epub 2018 Aug 16. PMID 30170779
- [Background] Olveira G, Tapia MJ, Ocon J, Cabrejas-Gomez C, Ballesteros-Pomar MD, Vidal-Casariego A, Arraiza-Irigoyen C, Olivares J, Conde-Garcia MC, Garcia-Manzanares A, Botella-Romero F, Quilez-Toboso RP, Matia P, Rubio MA, Chicharro L, Burgos R, Pujante P, Ferrer M, Zugasti A, Petrina E, Manjon L, Dieguez M, Carrera MJ, Vila-Bundo A, Urgeles JR, Aragon-Valera C, Sanchez-Vilar O, Breton I, Garcia-Peris P, Munoz-Garach A, Marquez E, Del Olmo D, Pereira JL, Tous MC. Hypoglycemia in noncritically ill patients receiving total parenteral nutrition: a multicenter study. (Study group on the problem of hyperglycemia in parenteral nutrition; Nutrition area of the Spanish Society of Endocrinology and Nutrition). Nutrition. 2015 Jan;31(1):58-63. doi: 10.1016/j.nut.2014.04.023. Epub 2014 May 10. PMID 25441588
- [Background] Feng Y, Barrett M, Hou Y, Yoon HK, Ochi T, Teitelbaum DH. Homeostasis alteration within small intestinal mucosa after acute enteral refeeding in total parenteral nutrition mouse model. Am J Physiol Gastrointest Liver Physiol. 2016 Feb 15;310(4):G273-84. doi: 10.1152/ajpgi.00335.2015. Epub 2015 Dec 3. PMID 26635320
- [Background] Pironi L, Steiger E, Joly F, Jeppesen PB, Wanten G, Sasdelli AS, Chambrier C, Aimasso U, Mundi MS, Szczepanek K, Jukes A, Theilla M, Kunecki M, Daniels J, Serlie M, Poullenot F, Cooper SC, Rasmussen HH, Compher C, Seguy D, Crivelli A, Santarpia L, Guglielmi FW, Kozjek NR, Schneider SM, Ellegard L, Thibault R, Matras P, Matysiak K, Van Gossum A, Forbes A, Wyer N, Taus M, Virgili NM, O'Callaghan M, Chapman B, Osland E, Cuerda C, Udvarhelyi G, Jones L, Won Lee AD, Masconale L, Orlandoni P, Spaggiari C, Diez MB, Doitchinova-Simeonova M, Serralde-Zuniga AE, Olveira G, Krznaric Z, Czako L, Kekstas G, Sanz-Paris A, Jauregui MEP, Murillo AZ, Schafer E, Arends J, Suarez-Llanos JP, Youssef NN, Brillanti G, Nardi E, Lal S; Home Artificial Nutrition and Chronic Intestinal Failure Special Interest Group of ESPEN; European Society for Clinical Nutrition and Metabolism. Characteristics of adult patients with chronic intestinal failure due to short bowel syndrome: An international multicenter survey. Clin Nutr ESPEN. 2021 Oct;45:433-441. doi: 10.1016/j.clnesp.2021.07.004. Epub 2021 Jul 28. PMID 34620351
- [Background] Derenski K, Catlin J, Allen L. Parenteral Nutrition Basics for the Clinician Caring for the Adult Patient. Nutr Clin Pract. 2016 Oct;31(5):578-95. doi: 10.1177/0884533616657650. Epub 2016 Jul 20. PMID 27440772
- [Background] Pironi L, Cuerda C, Jeppesen PB, Joly F, Jonkers C, Krznaric Z, Lal S, Lamprecht G, Lichota M, Mundi MS, Schneider SM, Szczepanek K, Van Gossum A, Wanten G, Wheatley C, Weimann A. ESPEN guideline on chronic intestinal failure in adults - Update 2023. Clin Nutr. 2023 Oct;42(10):1940-2021. doi: 10.1016/j.clnu.2023.07.019. Epub 2023 Jul 29. PMID 37639741
- [Background] Pironi L, Boeykens K, Bozzetti F, Joly F, Klek S, Lal S, Lichota M, Muhlebach S, Van Gossum A, Wanten G, Wheatley C, Bischoff SC. ESPEN practical guideline: Home parenteral nutrition. Clin Nutr. 2023 Mar;42(3):411-430. doi: 10.1016/j.clnu.2022.12.003. Epub 2023 Jan 9. PMID 36796121